CLINICAL TRIAL: NCT05355597
Title: "The Efficacy of Exparel Versus a Multidrug Cocktail in Soft Tissue Tumors"
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Physician left institution
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, James Wittig, Dr., Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1429450
Record Dates: First submitted 2022-04-07; First posted 2022-05-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Diseases; Soft Tissue Mass
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Epinephrine; Clonidine

STUDY DESIGN:
Intervention Model Description: Total of 140 subjects are recruited. Group A Receives one drug (70) and Group B receives the other drug (70)
Who Masked: Participant, Care Provider
Masking Description: This a double blinded study in which the investigator nor subjects will know which drug he or she receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel Group (Experimental): 70 subjects will receive Exparel
  Interventions: Drug: Exparel Injectable Product
- Multi-Drug Cocktail Group (Experimental): 70 subjects will receive a Multi-drug Cocktail
  Interventions: Drug: Multi-Drug Cocktail (Ropivicaine, Epinephrine, Ketolorac, Clonidine)

INTERVENTIONS:
Drug: Exparel Injectable Product — Both drugs have same desired effect. Will be injected intra-operatively while subjects are under anesthesia to alleviate significant post-operative pain.
  Arms: Exparel Group
Drug: Multi-Drug Cocktail (Ropivicaine, Epinephrine, Ketolorac, Clonidine) — Same desired effect as Exparel but different mechanism of action. Will be injected intra-operatively while subjects are under anesthesia to alleviate significant post-operative pain.
  Arms: Multi-Drug Cocktail Group

SUMMARY:
The objective of this proposed project is to determine which local anesthetic is more efficacious for use in soft tissue tumors: Exparel (liposomal bupivacaine) or a cocktail of Ropivicaine, Epinepherine, Ketolorac and Clonidine. This study will examine patients' post-operative pain levels as well as their narcotic consumption after removal of a soft tissue tumor while hospitalized and then twice daily through postoperative day 14.

DETAILED DESCRIPTION:
In recent years, there has been a substantial push to create a post-surgical protocol consisting of multimodal analgesia across multiple surgical subspecialties to decrease narcotic consumption and cost1. The negative side effects of narcotics and their addiction potential are well understood.

One of the modes of analgesia currently in use to mitigate surgical pain is some form of local anesthetic. Increasing the duration of analgesia has been sought after since its inception. Subsequently, longer acting anesthetics like bupivacaine have been implemented as well as supplementing their use with other drugs, such as epinephrine, to increase their effect duration and overall efficacy2. This has led to the development of Liposomal Bupivicaine or Exparel (TM, Parsippany NJ etc.) Exparel works by infusing liposomes in the administration of the long acting local analgesic which entrap the biologically active drug and slowly release it over a period of 72-96 hours 3-4. Thus, post-operative pain can be managed via direct injection of the drug at the surgical site with upwards to four days of pain relief.

Exparel has been studied extensively in the surgical literature; although within orthopedics, it has been primarily in regard to arthroplasty5. There has yet to be a study to illicit the best form of post-operative pain control in the world of orthopedic oncology, specifically in soft tissue tumors.

The objective of this proposed project is to determine which local anesthetic is more efficacious for use in soft tissue tumors: Exparel (liposomal bupivacaine) or a cocktail of Ropivicaine, Epinepherine, Ketolorac and Clonidine. This study will examine patients' post-operative pain levels as well as their narcotic consumption after removal of a soft tissue tumor while hospitalized and then twice daily through postoperative day 14.

ELIGIBILITY:
Inclusion Criteria:

* All primary soft tissue tumors
* Any adult patient (over 18 years old) with a soft tissue tumor confirmed with advanced imaging.

Two different study groups will be examined:

* Those patients undergoing resection of their soft tissue tumor intraoperatively injected with Exparel
* Those patients undergoing resection of their soft tissue tumor intraoperatively injected with the cocktail.
* Those two groups will be further stratified by anatomic location; Upper vs lower extremity, size; tumors ≥ 10cm, tumors ≥ 5cm, tumors < 5cm, and depth; superficial vs deep.

Exclusion Criteria:

* Pediatric Patients
* Patients without soft tissue tumors
* Tylenol or oxycodone allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Pain Outcomes | 14 days
  Pain will be recorded on a sheet for each patient. Self-reported, patient will describe pain each day on a scale of 1-10 (10 being the worst)

SECONDARY OUTCOMES:
Medication Consumption | 14 days
  Patient will self-report how much medication he or she took each day post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers, but we do anticipate publishing the results in a journal.

REFERENCES:
- [Background] Kelly MA. Current Postoperative Pain Management Protocols Contribute to the Opioid Epidemic in the United States. Am J Orthop (Belle Mead NJ). 2015 Oct;44(10 Suppl):S5-8. PMID 26447431
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Ranade VV. Drug delivery systems. 1. site-specific drug delivery using liposomes as carriers. J Clin Pharmacol. 1989 Aug;29(8):685-94. doi: 10.1002/j.1552-4604.1989.tb03403.x. PMID 2674208
- [Background] Barrington JW. Efficacy of Periarticular Injection With a Long-Acting Local Analgesic in Joint Arthroplasty. Am J Orthop (Belle Mead NJ). 2015 Oct;44(10 Suppl):S13-6. PMID 26447426